## MECHANISMS AND PHENOTYPES OF HYPERTENSION IN PATIENTS IN CHRONIC HEMODIALYSIS

NCT06764277

DATE: 09/11/2025

STATISTICAL ANALYSES

## Statistical analyses.

All statistical analyses will be performed using GraphPad Prism version 10. The normality of data distributions was assessed using the Kolmogorov–Smirnov test. For comparisons between two groups, unpaired Student's t-tests will be applied when data followed a normal distribution, and the Mann–Whitney U test will be used for non-normally distributed data. For comparisons among more than two groups, one-way analysis of variance (ANOVA) will be performed for normally distributed data, followed by Tukey's post hoc test. When data did not meet normality assumptions, the Kruskal–Wallis test will be used, followed by Dunn's post hoc test for multiple comparisons.

For all analyses, two-tailed p-values < 0.05 will be considered statistically significant. The assumptions underlying parametric tests (normality and homogeneity of variances) will be verified prior to analysis; if assumptions were not met, appropriate non-parametric alternatives will be used as described above.